CLINICAL TRIAL: NCT02549001
Title: A Multicenter, Randomized, Double-blind, Parallel, Vehicle-controlled Study to Evaluate the Efficacy and Safety of P-3058 10% Nail Solution in the Treatment of Onychomycosis
Brief Title: Study to Evaluate the Efficacy and Safety of P-3058 10% Nail Solution in the Treatment of Toenail Onychomycosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polichem S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PM1331; 2015-000561-31 (EudraCT Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Nail fungus
MeSH Terms: conditions — Onychomycosis | interventions — amorolfine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- P-3058 10% (Experimental): P-3058 10%
  Interventions: Drug: P-3058 10%
- vehicle of P-3058 10% (Placebo Comparator): vehicle of P-3058 10%
  Interventions: Drug: vehicle of P-3058 10%
- amorolfine 5% (Active Comparator): Loceryl®
  Interventions: Drug: amorolfine 5%

INTERVENTIONS:
Drug: P-3058 10%
  Arms: P-3058 10%
Drug: vehicle of P-3058 10%
  Arms: vehicle of P-3058 10%
Drug: amorolfine 5%
  Other Names: Loceryl®
  Arms: amorolfine 5%

SUMMARY:
The purpose of this study is to determine whether P-3058 nail solution is a safe and effective treatment for onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients aged 12 years and older of any race.
* Males or females.
* Patients with onychomycosis involving ≥ 20% to ≤ 50% of target big toenail.
* Patients with a positive KOH examination and culture positive for dermatophyte

Exclusion Criteria:

* Presence of "yellow spikes" on the target nail.
* Presence of dermatophytoma on the target nail.
* Presence of nail thickness exceeding 2 mm.
* Patients with proximal subungual involvement
* Patients with severe plantar or moccasin tinea pedis
* Patients with nail abnormalities due to other conditions
* Patients with life expectancy less than 2 years.
* Chemotherapy, immunosuppressive therapy in the 12 weeks prior to Screening visit (V1).
* Systemic corticosteroids, antimetabolites and immune-stimulants therapy in the 4 weeks prior to Screening visit (V1).
* HIV infection or any other immunodeficiency.
* Alcohol or substance abuse.
* Patients with history of allergic reactions to terbinafine or its excipients.
* Woman who is pregnant, nursing an infant, or planning a pregnancy during the study period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 953 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Complete cure of target great toenail defined as negative KOH microscopy, negative culture for dermatophytes and target nail totally clear. | Week 60

SECONDARY OUTCOMES:
Responder rate of the target toenail, defined as negative KOH microscopy, negative culture for dermatophytes and ≤10% residual involvement of the target toenail. | Week 60
Negative culture rate for dermatophytes of the target nail. | Week 60
Mycological cure defined as negative KOH microscopy and negative culture for dermatophytes of the target nail. | Week 60
Overall safety by recording any AE during the entire study duration and the local tolerability by means of severity scores for skin irritation. | Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Caserini, MD, Study Director — Polichem S.A.
Locations (13):
- Polichem Investigative Site, Multiple Locations, Belgium
- Polichem Investigative Site, Multiple Locations, Bulgaria
- Polichem Investigative Site, Multiple Locations, Czechia
- Polichem Investigative Site, Multiple Locations, Germany
- Polichem Investigative Site, Multiple Locations, Greece
- Polichem Investigative Site, Multiple Locations, Hungary
- Polichem Investigative Site, Various Cities in Iceland, Iceland
- Polichem Investigative Site, Multiple Locations, Latvia
- Polichem Investigative Site, Multiple Locations, Lithuania
- Polichem Investigative Site, Multiple Locations, Poland
- Polichem Investigative Site, Multiple Locations, Russia
- Polichem Investigative Site, Multiple Locations, Slovakia
- Polichem Investigative Site, Multiple Locations, Sweden